CLINICAL TRIAL: NCT02415712
Title: Specified Drug-use Survey of Fomepizole Intravenous Infusion "Takeda" (All-case Surveillance)
Brief Title: Specified Drug-use Survey of Fomepizole Intravenous Infusion (All-case Surveillance)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Fomepizole-5001; jRCT1080222765 (Registry Identifier: jRCT)
Record Dates: First submitted 2015-03-24; First posted 2015-04-14 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Ethylene Glycol Poisoning, Methanol Poisoning
Keywords: Pharmacotherapy
MeSH Terms: interventions — Fomepizole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fomepizole Intravenous Infusion: Fomepizole Intravenous Infusion
  Interventions: Drug: Fomepizole

INTERVENTIONS:
Drug: Fomepizole — The first dose of fomepizole is administered at a dose of 15 mg/kg, followed by the second to fifth doses administered at a dose of 10 mg/kg. The sixth and subsequent doses are administered at a dose of 15 mg/kg. The interval of the intravenous doses is 12 hours with one administration lasting more than 30 minutes.
  Other Names: Fomepizole Intravenous Infusion 1.5 g

SUMMARY:
The objective of this survey is to evaluate the safety and efficacy of fomepizole intravenous infusion in Japanese patients with ethylene glycol and methanol poisonings in daily medical practice.

DETAILED DESCRIPTION:
Clinical studies for fomepizole intravenous infusion have not been conducted in Japan, and there are few reports of data on drug-use, including in the literature, in Japanese patients; therefore, an evaluation of the safety and efficacy of fomepizole intravenous infusion is required.

This specified drug-use survey for fomepizole intravenous infusion (Fomepizole Intravenous Infusion 1.5 g "Takeda," hereinafter referred to as "the drug") was planned to evaluate the safety and efficacy of the drug in patients with ethylene glycol and methanol poisoning in daily medical practice.

ELIGIBILITY:
Inclusion Criteria:

-All patients who have been confirmed as receiving the drug

Exclusion Criteria:

-None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ethylene glycol poisoning or methanol poisoning
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Takeda Sponsored Site, Osaka
  - Takeda Sponsored Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60234db2bf003ab496e5

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 91 investigative sites in Japan, from 27 January 2015 to 30 June 2022.
Pre-assignment Details: Participants with a historical diagnosis of ethylene glycol and methanol poisonings were enrolled. Participants received fomepizole as part of a routine medical care.
Groups:
- Fomepizole Intravenous Infusion: The first dose of fomepizole is administered at a dose of 15 mg/kg, followed by the second to fifth doses administered at a dose of 10 mg/kg. The sixth and subsequent doses are administered at a dose of 15 mg/kg. The interval of the intravenous doses is 12 hours with one administration lasting more than 30 minutes.
Period: Overall Study
Arm/Group | Fomepizole Intravenous Infusion
Started | 147
Completed | 131
Not Completed | 16
Not completed — Protocol Violation | 16

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Fomepizole Intravenous Infusion
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 130
    (all) | 43.6 (20.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 87
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 131
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — Number of participants who had or did not have a liability or tendency to suffer from hypersensitivity was reported. Unknown: Data could not be collected.
  Participants
    Had No Predisposition to Hypersensitivity | 108
    Had Predisposition to Hypersensitivity | 11
    Unknown | 12
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above. Unknown: Data could not be collected.
  Participants
    Had No Medical Complications | 52
    Had Medical Complications | 78
    Unknown | 1
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above. Unknown: Data could not be collected.
  Participants
    Had No Medical History | 94
    Had Medical History | 33
    Unknown | 4
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 115
    (all) | 162.9 (14.01)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 123
    (all) | 60.99 (16.752)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2
    number analyzed (Participants) | 115
    (all) | 22.71 (4.780)
Alcohol Consumption (at Time of Poisoning) [Count of Participants; unit: Participants] — Number of participants who had been consuming alcohol at the time of poisoning was reported. Unknown: Data could not be collected.
  Participants
    No | 80
    Yes | 27
    Unknown | 24
Pregnancy Status [Count of Participants; unit: Participants] — This baseline characteristic was analyzed only in female participants. Unknown: Data could not be collected. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 44
    Not Pregnant | 42
    Pregnant | 0
    Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: From the first dose to 24 hours after the last dose of the drug (Up to approximately 11 days)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Fomepizole Intravenous Infusion
Number analyzed (Participants) | 131
Participants | 22

2. Primary Outcome: Number of Participants Who Had One or More Adverse Drug Reactions
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.
Time Frame: From the first dose to 24 hours after the last dose of the drug (Up to approximately 11 days)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Fomepizole Intravenous Infusion
Number analyzed (Participants) | 131
Participants | 7

3. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Events (SAEs)
Description: A serious AE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: From the first dose to 24 hours after the last dose of the drug (Up to approximately 11 days)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Fomepizole Intravenous Infusion
Number analyzed (Participants) | 131
Participants | 13

4. Primary Outcome: Number of Participants Who Had One or More Serious Adverse Drug Reactions
Description: A serious AE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Serious adverse drug reaction refers to serious AE that are related to administered drug.
Time Frame: From the first dose to 24 hours after the last dose of the drug (Up to approximately 11 days)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Fomepizole Intravenous Infusion
Number analyzed (Participants) | 131
Participants | 0

5. Primary Outcome: Arterial Blood pH
Description: pH in arterial blood values at baseline, 4 hours after the first dose, and 24 hours after the last dose (Up to approximately 11 days) were reported.
Time Frame: Baseline, 4 hours after the first dose, and 24 hours after the last dose (Up to approximately 11 days)
Population: Participants in the Efficacy Analysis Set for whom test value/s from at least one assessment time point is/are available from both before and after the start of fomepizole intravenous infusion.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Fomepizole Intravenous Infusion
Number analyzed (Participants) | 91
pH
  Baseline | 7.3010 (0.16064)
  4 Hours after the First Dose: number analyzed (Participants) | 58
  4 Hours after the First Dose | 7.4042 (0.06809)
  24 Hours after the Last Dose: number analyzed (Participants) | 42
  24 Hours after the Last Dose | 7.4120 (0.05078)

ADVERSE EVENTS:
Time Frame: From the first dose to 24 hours after the last dose of the drug (Up to approximately 11 days)
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Fomepizole Intravenous Infusion
All-Cause Mortality (participants affected / at risk) | 7/131
Serious Adverse Events (participants affected / at risk) | 13/131
Other Adverse Events (participants affected / at risk) | 3/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fomepizole Intravenous Infusion (N=131)
Acidosis (Metabolism and nutrition disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Putamen haemorrhage (Nervous system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Death (General disorders) | 2 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Multiple organ dysfunction syndrome (General disorders) | 1
Blood pressure decreased (Investigations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fomepizole Intravenous Infusion (N=131)
Vomiting (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT02415712/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT02415712/SAP_001.pdf